CLINICAL TRIAL: NCT00133900
Title: Circulating Tumor Cells and the Prediction of Overall Survival in Patients With Androgen Independent Prostate Cancer Entering Onto Chemotherapy
Brief Title: Circulating Tumor Cells and Survival in Hormone Refractory Prostate Cancer (HRPC) Patients Receiving Chemotherapy
Acronym: IMMC-38
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Immunicon (Industry)
Responsible Party: Senior Director, Clinical Development, Immunicon
Other Study IDs: IMMC-38
Record Dates: First submitted 2005-08-22; First posted 2005-08-24 (Estimated); Last update posted 2009-07-28 (Estimated); Status verified 2008-03

CONDITIONS: Hormone Refractory Prostate Cancer; Prostate Cancer
Keywords: hormone refractory prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Phlebotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum Samples and RNA samples have been retained.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort: Metastatic Hormone Refractory Prostate Cancer Patients
  Interventions: Procedure: Phlebotomy

INTERVENTIONS:
Procedure: Phlebotomy — Peripheral blood draws for evaluation of circulating tumor cells

SUMMARY:
This study enrolled men with prostate cancer who had failed hormone therapy (as shown by rising prostate-specific antigen [PSA] levels) and who were about to start a new line of chemotherapy. Blood was drawn prior to the patient receiving chemotherapy and then monthly thereafter for up to 18 months or until disease progression, whichever occurred first. The blood was tested to find circulating tumor cells (CTC) and to count them. The circulating tumor cell levels were studied in relation to the patient's overall survival. Serum was also collected for PSA testing, and additional blood samples were drawn to test for circulating endothelial cells and RNA was isolated for future gene expression testing.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 18 years
* Pathological diagnosis of adenocarcinoma of the prostate
* First or later line of chemotherapy
* Serum testosterone < 50ng/mL
* ECOG 0-2
* Serum PSA > or = 5ng/mL
* PSA progression (2 rises above a reference value)
* Bone scan within 60 days of enrollment
* Computed tomography (CT) scan
* If measurable disease, bone scans every 6-8 months

Exclusion Criteria:

* Systemic radiation
* Prior history of other carcinoma within the last 5 years, except non-melanoma skin cancer
* Brain metastases

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Oncology patients from academic institutions and private practices
Sampling Method: Probability Sample
Enrollment: 276 (Actual)
Dates: Start 2004-12; Primary Completion 2009-02 (Estimated); Study Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Up to 36 months from time of baseline draw

SECONDARY OUTCOMES:
Progression Free Survival | Up to 36 months after baseline draw

CONTACTS AND LOCATIONS:
Overall Officials: Ken Pienta, MD, Principal Investigator — University of Michigan; Derek Raghavan, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Coumans FA, Ligthart ST, Uhr JW, Terstappen LW. Challenges in the enumeration and phenotyping of CTC. Clin Cancer Res. 2012 Oct 15;18(20):5711-8. doi: 10.1158/1078-0432.CCR-12-1585. Epub 2012 Sep 25. PMID 23014524
- See also: 510(k) Premarket Notification Summary — http://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfPMN/pmn.cfm?ID=22145